CLINICAL TRIAL: NCT05861895
Title: A Multi-Regional, Open-Label, Dose Escalation and Dose Expansion Phase Ⅰ Clinical Study to Investigate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of HF158K1 in Participants With HER-2 Positive or HER-2 Low Expression Advanced Solid Tumors
Brief Title: A Clinical Study to Investigate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of HF158K1 in Participants With HER-2 Positive or HER-2 Low Expression Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HighField Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HF158K1-101
Record Dates: First submitted 2023-04-20; First posted 2023-05-17 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Solid Tumors, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dose escalation cohort 1: HF158K1 given Q3W at 2 mg/m² (Experimental): Participants in this dose group(2 mg/m²) will receive HF158K1 on D1 of each treatment cycle (3 weeks as a treatment cycle) through intravenous infusion.
  Interventions: Drug: HF158K1 /Arm 2 mg/m²
- Dose escalation cohort 1: HF158K1 given Q3W at 6 mg/m² (Experimental): Participants in this dose group(6 mg/m²) will receive HF158K1 on D1 of each treatment cycle (3 weeks as a treatment cycle) through intravenous infusion.
  Interventions: Drug: HF158K1 /Arm 6 mg/m²
- Dose escalation cohort 1: HF158K1 given Q3W at 15 mg/m² (Experimental): Participants in this dose group(15 mg/m²) will receive HF158K1 on D1 of each treatment cycle (3 weeks as a treatment cycle) through intravenous infusion.
  Interventions: Drug: HF158K1 /Arm 15 mg/m²
- Dose escalation cohort 1: HF158K1 given Q3W at 30 mg/m² (Experimental): Participants in this dose group(30 mg/m²) will receive HF158K1 on D1 of each treatment cycle (3 weeks as a treatment cycle) through intravenous infusion.
  Interventions: Drug: HF158K1 /Arm 30 mg/m²
- Dose escalation cohort 1: HF158K1 given Q3W at 45 mg/m² (Experimental): Participants in this dose group(45 mg/m²) will receive HF158K1 on D1 of each treatment cycle (3 weeks as a treatment cycle) through intravenous infusion.
  Interventions: Drug: HF158K1 /Arm 45 mg/m²
- Dose escalation cohort 1: HF158K1 given Q3W at 60 mg/m² (Experimental): Participants in this dose group(60 mg/m²) will receive HF158K1 on D1 of each treatment cycle (3 weeks as a treatment cycle) through intravenous infusion.
  Interventions: Drug: HF158K1 /Arm 60 mg/m²

INTERVENTIONS:
Drug: HF158K1 /Arm 2 mg/m² — Duration of infusion: HF158K1 is diluted using 5% (50 mg/ml) glucose injection or 0.9% sodium chloride injection (saline) to a total volume of 250 ml and is administered through intravenous infusion for 90 ± 10 min.
  Other Names: Infusion
  Arms: Dose escalation cohort 1: HF158K1 given Q3W at 2 mg/m²
Drug: HF158K1 /Arm 6 mg/m² — Duration of infusion: HF158K1 is diluted using 5% (50 mg/ml) glucose injection or 0.9% sodium chloride injection (saline) to a total volume of 250 ml and is administered through intravenous infusion for 90 ± 10 min.
  Other Names: Infusion
  Arms: Dose escalation cohort 1: HF158K1 given Q3W at 6 mg/m²
Drug: HF158K1 /Arm 15 mg/m² — Duration of infusion: HF158K1 is diluted using 5% (50 mg/ml) glucose injection or 0.9% sodium chloride injection (saline) to a total volume of 250 ml and is administered through intravenous infusion for 90 ± 10 min.
  Other Names: Infusion
  Arms: Dose escalation cohort 1: HF158K1 given Q3W at 15 mg/m²
Drug: HF158K1 /Arm 30 mg/m² — Duration of infusion: HF158K1 is diluted using 5% (50 mg/ml) glucose injection or 0.9% sodium chloride injection (saline) to a total volume of 250 ml and is administered through intravenous infusion for 90 ± 10 min.
  Other Names: Infusion
  Arms: Dose escalation cohort 1: HF158K1 given Q3W at 30 mg/m²
Drug: HF158K1 /Arm 45 mg/m² — Duration of infusion: HF158K1 is diluted using 5% (50 mg/ml) glucose injection or 0.9% sodium chloride injection (saline) to a total volume of 250 ml and is administered through intravenous infusion for 90 ± 10 min.
  Other Names: Infusion
  Arms: Dose escalation cohort 1: HF158K1 given Q3W at 45 mg/m²
Drug: HF158K1 /Arm 60 mg/m² — Duration of infusion: HF158K1 is diluted using 5% (50 mg/ml) glucose injection or 0.9% sodium chloride injection (saline) to a total volume of 250 ml and is administered through intravenous infusion for 90 ± 10 min.
  Other Names: Infusion
  Arms: Dose escalation cohort 1: HF158K1 given Q3W at 60 mg/m²

SUMMARY:
HF158K1 is an investigational liposome form of doxorubicin hydrochloride, an anthracycline topoisomerase inhibitor, encapsulated by lipid membranes containing TL01, a HER2-directed Trastuzumab Fab fragment conjugated lipid.

DETAILED DESCRIPTION:
This study is a multi-regional, open-label, multiple-dose administration dose-escalation and dose-expansion study, including a Dose-Escalation Phase (Ia) and a Dose-Expansion Phase (Ib).

HF158K1 contains multiple copies of the targeting antibody on liposome surface. It is designed to bind and deliver the chemotherapeutic doxorubicin to tumor cells at even very low HER2 expression levels. The study recruits patients with unresectable or metastatic advanced solid tumors (HER-2 positive (IHC 3+, or IHC 2+ with ISH +) or HER-2 low expression (IHC 2+ with ISH -, or IHC 1+)) who have failed or are intolerant (disease progression, or intolerance to chemotherapy, targeted therapy, etc.) to standard treatment, or currently have no available treatment regimen.

Phase 1a(Dose escalation) will assess the safety，tolerability，pharmacokinetics of HF158K1 in participants to determine the maximum tolerated dose (MTD) of HF158K1 through the incidence of dose-limiting toxicity (DLT).

Phase 1b(Dose expansion) will assess safety and preliminary efficacy of HF158K1 in participants with specific tumor types in selected dose groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntary to participate in the clinical study, sign a written informed consent form, and able to comply with clinical visits and study-related procedures.

  2. Male or female participants at least 18 years old when signing the informed consent form.

  3. ECOG performance score of 0 to 1 point. 4. Study population: HER-2 positive (IHC 3+, or IHC 2+ with ISH +) or HER-2 low expression (IHC 2+ with ISH -, or IHC 1+) participants with unresectable or metastatic advanced solid tumors (confirmed by histopathology or cytology analysis) who have failed or are intolerant (disease progression, or intolerance to chemotherapy, targeted therapy, etc.) to standard treatment, or currently have no available treatment regimen.

  5. Expected survival of at least 3 months. 6. According to the RECIST v1.1 criteria, there is at least one measurable lesion in the dose expansion stage.

  7. The functional level of bone marrow reserve and organs must meet the following requirements (without ongoing continuous supportive treatment): Bone marrow reserve: neutrophil count (NE#) ≥ 1.5×109/L, platelet count (PLT) ≥ 90×109/L, and hemoglobin (HGB) > 9.0 g/dL (no blood transfusion or hematopoietic stimulating factor therapy within 14 days).

Coagulation function: activated partial prothrombin time (APTT) prolonged to ≤1.5×ULN, and international normalized ratio (INR) ≤1.5.

Liver function: total bilirubin (TBIL) ≤ 1.5×ULN, and alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 2.5×ULN, if there is liver metastasis, ALT and AST ≤ 5×ULN and TBIL≤ 3×ULN.

Renal function: creatinine clearance ≥ 50 mL/min or serum creatinine ≤ 1.5×ULN. 8. Eligible Participants with fertility (male and female) must agree to use reliable contraceptive methods with their partners and have no plan to have baby during the study period and at least 6 months after the last administration. female Participants of childbearing age must have a negative serum or urine pregnancy test during screening period and before the first dose.

9. Other participants that can potentially benefit from the investigational drug as assessed by the investigator.

Exclusion Criteria:

* 1. Participants who are known to be allergic to doxorubicin and/or other similar compounds, or to any of excipients of HF158K1, or participants with allergic constitution (multiple drug and food allergies).

  2. Participants who have used doxorubicin prior to screening with a total cumulative dose > 350 mg/m2 (other anthracyclines converted by 1 mg doxorubicin equivalence: 2 mg epirubicin, or 2 mg epirubicin, or 2 mg zolpidem, or 0.5 mg demethoxyzolpidem), or who have received anthracyclines and suffered severe cardiotoxicity, or who discontinued doxorubicin liposome therapy due to serious adverse events.

  3. Participants who received radiotherapy or chemotherapy (paclitaxel, cyclosporine, dextropropylenol, cytarabine, streptozotocin, etc.) within 4 weeks prior to first dose administration, or received other antitumor therapy such as endocrine therapy, herbal therapy, or local radiation therapy for pain relief within 2 weeks prior to first dose administration, except for the following: Nitrosourea or mitomycin C within 6 weeks prior to the first administration of the investigational drug.

Oral fluorouracil-based and small-molecule targeted drugs for 2 weeks prior to the first administration of the investigational drug or within 5 half-lives of the drug (whichever is longer).

4. Participants with brain parenchymal metastases or meningeal metastases with clinical symptoms that, in the judgment of the investigator, are not suitable for enrollment (those who have received prior treatment (radiation or surgery) for systemic, radical brain metastases, have maintained imaging- confirmed stability for at least 28 days, and have discontinued systemic steroid therapy for > 14 days without clinical symptoms will be allowed for enrollment).

5. Participants who have not recovered to < Grade 1 (according to CTCAE 5.0) or to pre-treatment baseline levels from all prior treatment-induced adverse events prior to the first dose (except for adverse events without safety risks as judged by the investigator, such as alopecia, Grade 2 peripheral neurotoxicity, and stabilized hypothyroidism under hormone replacement therapy).

6. Participants who are taking (or are not able to discontinue until at least 1 week before the first dose of the study) any drug known to strongly inhibit or strongly induce CYP3A4, CYP2D6 or P-gp.

7. Participants with a history of serious cardiovascular and cerebrovascular diseases, including but not limited to: Serious heart rhythm or conduction abnormalities, such as ventricular arrhythmia that requires clinical intervention, degree II-III atrioventricular block, etc.

Cardiac function: left ventricular ejection fraction (LVEF) ≤ 50%, corrected QT interval (QTcF) > 470 ms.

Thromboembolic events requiring therapeutic anticoagulation within 3 months before the first administration, or participants with venous filters.

Participants with Class III~IV cardiac insufficiency according to the New York Heart Association (NYHA) criteria.

Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other Grade 3 and above cardiovascular and cerebrovascular events within 6 months before the first administration.

Clinically uncontrollable hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg), and patients with a history of hypertension were allowed to enroll as long as their blood pressure was controlled below this limitation through antihypertensive therapy.

Any factors that increase the risk of QTc prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, or use of any concomitant drug that are known to or may prolong the QT interval.

8. Participants who have received last dose of any other investigational drug product or treatments within 28 days prior to the first administration of the investigational drug.

9. Participants who have undergone major organ surgery (excluding needle biopsy，tracheotomy, gastrostomy, etc.) or had significant trauma within 28 days before the first administration of investigational drug or need to undergo elective surgery during the study period.

10. Participants with a serious unhealable wound/ulcer/fracture within 28 days before the first administration of the investigational drug.

11. Participants with an active infection within 1 week prior to the first administration of the investigational drug and currently require intravenous anti-infection therapy.

12. Third space effusion that cannot be clinically controlled and is not suitable for enrollment as judged by the investigator.

13. Known history of drug abuse. 14. Participants with mental disorders or poor compliance. 15. HIV infection, active HBV infection (HBV DNA > ULN), or active HCV infection (HCV RNA > ULN).

16. Women who are pregnant or breastfeeding. 17. Participants who cannot tolerate venous blood sampling. 18. The investigator believes that the participant has a history of other serious systemic diseases or is not suitable for participating in this clinical study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-04-23 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | The period of AE collection starts after the participant receives the investigational drug, until 28±3 days after the EOT/early withdrawal or before the participant starts another anti-tumor treatment (whichever occurs first).
  Defined by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE V5.0)
Incidence of dose-limiting toxicities(DLT) | The DLT evaluation period is from the first administration of the investigational drug to the end of the first treatment cycle, lasting for 21 days.（only Ia）
  Observe the dose limiting toxicity, and Incidence of dose-limiting toxicities(DLT) will be assessed
Red blood cell count in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Red blood cell count in whole blood
White blood cell in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for white blood cell count in whole blood
Hematocrit in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Hematocrit in whole blood
Neutrophil count in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for neutrophil count in whole blood
Hemoglobin concentration in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for hemoglobin concentration in whole blood
Percentage of lymphocytes (LYM%) | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Percentage of lymphocytes (LYM%) in whole blood
Lymphocyte count | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Lymphocyte count in whole blood
Percentage of neutrophils (NEU%) Percentage of neutrophils (NEU%) | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Percentage of neutrophils (NEU%) in whole blood
Platelet count in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Platelet count in whole blood
Prothrombin time in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Prothrombin time in whole blood sample
International normalized ratio in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for international standardized ratio in whole blood sample
Fibrinogen in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Fibrinogen in whole blood
Activated partial prothrombin time in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for activated partial thromboplastin time in whole blood sample
Total bilirubin concentration in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for total bilirubin concentration in whole blood sample
ALT concentration in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for alanine aminotransferase(ALT) concentration in whole blood sample
AST concentration in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for aspartate aminotransferase(AST) concentration in whole blood sample
Total protein concentration in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for total protein concentration in whole blood sample
Urea concentration in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for urea concentration in whole blood sample
Creatinine concentration in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for creatinine concentration in whole blood sample
Total cholesterol concentration in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for total cholesterol concentration in whole blood sample
Triglycerides concentration in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for triglycerides concentration in whole blood sample
HDL-C in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for high density lipoprotein cholesterol (HDL-C) in whole blood sample
LDL-C in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for low density lipoprotein cholesterol (LDL-C) in whole blood sample
Glucose in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Lactic dehydrogenase in whole blood
Alkaline phosphatase in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Lactic dehydrogenase in whole blood
Lactic dehydrogenase in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Lactic dehydrogenase in whole blood
Gamma-glutamyl transferase in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Gamma-glutamyl transferase in whole blood
Albumin in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Albumin in whole blood
Direct bilirubin in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Direct bilirubin in whole blood
Sodium in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Sodium in whole blood
Potassium in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Potassium in whole blood
Chloride in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Chloride in whole blood
Calcium in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Calcium in whole blood
Phosphate in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Phosphate in whole blood
Uric acid in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Uric acid in whole blood
Creatine kinase in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Creatine kinase in whole blood
Creatine kinase isoenzyme in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Creatine kinase isoenzyme in whole blood
Troponin-T (TnT) in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Troponin-T in whole blood
Troponin-I (TnI) in whole blood sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Troponin-I in whole blood
Urine protein in urine sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Urine protein in urine sample
Red blood cells in urine sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Red blood cells in urine sample
White blood cells in urine sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for White blood cells in urine sample
PH in urine sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for pH in urine sample
Ketone bodies in urine sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Ketone bodies in urine sample
Urine glucose in urine sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Urine glucose in urine sample
Urine bilirubin in urine sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Urine bilirubin in urine sample
Urine occult blood in urine sample | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Urine occult blood in urine sample
Heart Rate in beats per minute in beats per minute of ECG | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for heart rate in beats per minute
RR Interval by ECG | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for RR interval by ECG
PR Interval by ECG | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for PR interval by ECG
QRS Interval by ECG | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for QRS interval by ECG
QT Interval by ECG | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for QT interval by ECG
QTcF by ECG | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for QTcF interval by ECG
Left ventricular ejection fraction measured by Echocardiography | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Left ventricular ejection fraction measured by Echocardiography
Body (Ear) Temperature measurement in Vital Signs | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Body (Ear) Temperature
Pulse measurement in Vital Signs | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Pulse
Respiration Rate measurement in Vital Signs | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for respiration rate in breaths of Vital Signs
Sitting Systolic Blood Pressure | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Sitting Systolic Blood Pressure
Sitting Diastolic Blood Pressure | This should be evaluated during the screening period, on Day 1, 8, 15 of each cycle (each cycle is 21 days) , Day 1 of each subsequent cycle, at the EOT/early withdrawal and safety follow-up.
  Changes from baseline for Sitting Diastolic Blood Pressure
The recommended Phase II dose | After the end of the dose Expansion Phase（only Ib）
  Determine the Recommended Phase II Dose(mg/㎡) of HF158K1 and provide references for dose selection in future clinical studies.
Determine the maximum tolerated dose | The first administration of the investigational drug to the end of the first treatment cycle, lasting for 21 days.
  The dose at which the incidence of DLT was closest to the target probability of toxicity (30%).

SECONDARY OUTCOMES:
HF158K1 pharmacokinetic parameters with Cmax | Within 336 hours after the first and second administration
  Maximum plasma concentration (Cmax) after administration of HF158K1
AUC by plasma concentration of whole blood sample | Within 336 hours after the first and second administration
  Area under plasma concentration -time curve after dose
Tmax by plasma concentration of whole blood sample | Within 336 hours after the first and second administration
  Peak time (Tmax) after dose
T1/2 by plasma concentration of whole blood sample | Within 336 hours after the first and second administration
  Elimination half-life (T1/2) after dose
CL by plasma concentration of whole blood sample | Within 336 hours after the first and second administration
  Clearance (CL) after dose
Vd by plasma concentration of whole blood sample | Within 336 hours after the first and second administration
  Volume of distribution(Vd) after dose
AUClast by plasma concentration of whole blood sample | Within 336 hours after the first and second administration
  Ratios of geometric means of AUClast (Area under the plasma concentration-time curve from zero to time of last quantifiable concentration) after dose
The objective response rate(ORR) of HF158K1 | ORR will be calculated for all participants who have received the investigational drug at least once and have undergone at least one tumor evaluation after administration, assessed up to 51 weeks.
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR)
disease control rate (DCR) of HF158K1 | DCR will be calculated for all participants who have received the investigational drug at least once and have undergone at least one tumor evaluation after administration, assessed up to 51 weeks.
  DCR is defined as the proportion of participants with complete response stable disease and partial response (CR+PR+SD)
duration of response(DOR) of HF158K1 | DOR will be calculated for all participants who have received the investigational drug at least once and have undergone at least one tumor evaluation after administration, assessed up to 51 weeks.
  For duration of response (DOR), the Kaplan-Meier survival curve will be plotted to analyze their maximum, minimum, median and 95% confidence interval descriptively statistically.
Analysis of immunogenicity | On the first day of the first cycle, on the first day of the fourth cycle, on the 21st day of the eighth cycle
  Immunogenicity analyses related to anti-TL01 antibody will be performed based on IMS(Immunogenicity Analysis Set).

CONTACTS AND LOCATIONS:
Overall Officials: MINAL BARVE, Principal Investigator — Mary Crowley Cancer Research
Locations (1):
- Mary Crowley Cancer Research, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No